CLINICAL TRIAL: NCT06748950
Title: A Randomized Controlled Trial of a Ketogenic Metabolic Therapy in Schizophrenia, Bipolar Disorder, Major Depressive Disorder: Deep Omic Profiling
Brief Title: Ketogenic Metabolic Therapy in Schizophrenia, Bipolar Disorder, Major Depressive Disorder: Deep Omic Profiling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Shebani Sethi, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76425
Record Dates: First submitted 2024-12-14; First posted 2024-12-27 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia; Schizophrenia and Related Disorders; Bipolar Disorder; Bipolar and Related Disorders; Major Depressive Disorder; Major Depression Severe; Ketogenic Dieting; Ketosis; Metabolic Disease; Metabolic Syndrome
Keywords: Mental Illness; Multiomics; Multi-omics; Omics Profiling
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Bipolar and Related Disorders; Depressive Disorder, Major; Ketosis; Metabolic Diseases; Metabolic Syndrome; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Ketogenic Diet Only (Experimental): Participants will follow 12 weeks of the ketogenic diet, with monitoring of physical and psychological health and coaching support.
  Interventions: Other: LCHF Ketogenic Diet
- Arm 2: DAU- Ketogenic Diet Crossover (Experimental): Participants will follow 12 weeks of their usual diet (Diet-as-Usual, DAU). Then, participants will crossover and follow 12 weeks of the ketogenic diet. Monitoring of physical and psychological health and coaching support will occur throughout participation.
  Interventions: Other: LCHF Ketogenic Diet; Other: Diet-as-Usual (DAU)

INTERVENTIONS:
Other: LCHF Ketogenic Diet — Low Carbohydrate, Moderate Protein, High Fat (LCHF) Ketogenic Dietary Intervention for 12 weeks
Other: Diet-as-Usual (DAU) — Participant's usual diet
  Arms: Arm 2: DAU- Ketogenic Diet Crossover

SUMMARY:
The goal of this randomized clinical trial is to be adequately powered to evaluate the effect of ketogenic metabolic therapy on the quality of life in serious mental illness, schizophrenia, bipolar disorder, major depressive disorder.

DETAILED DESCRIPTION:
The ketogenic diet is a low carbohydrate, moderate protein, higher fat diet to help individuals improve energy and mood and to obtain nutrients from fats and protein. Schizophrenia, bipolar disorder, and major depressive disorder, collectively affect about 344 million individuals worldwide, (24 million with schizophrenia, 40 million people with BD, and 280 million with depression World Health Organization). These illnesses are debilitating psychiatric conditions characterized by a chronic pattern of emotional, behavioral, and cognitive disturbances. Shared psychopathology includes the pre-eminence of altered affective states, disorders of thoughts, and behavioral control. Additionally, those conditions share epidemiological traits, including significant cardiovascular, metabolic, infectious, and respiratory comorbidities, resulting in reduced life expectancy of up to 25 years (Xie et al., 2023). Reductions in cerebral glucose uptake are seen in both schizophrenia and bipolar disorder. While glucose is the brain's default fuel, ketone bodies are 27% more efficient, improve brain metabolism, and promote neural stability, as seen in childhood epilepsy (Sethi & Ford, 2022). The ketogenic diet (KD, also known as metabolic therapy) has been successful in the treatment of obesity, type 2 diabetes, and epilepsy (Sethi et al., 2024, Liu et al., 2018, Martin-McGill et al., 2020). Nutritional ketosis has been successfully used to treat a range of neurological disorders. Metabolic disorders, which include conditions such as obesity and metabolic syndrome, more commonly occur in individuals with severe mental illness (between 40-60%). The investigators aim to study the effect of ketogenic metabolic therapy on various markers including:

* Metabolic health measurements and cardiovascular risk factors including: insulin resistance, advanced lipid analysis, weight, glucose regulation, dyslipidemia, absolute body fat chang, inflammation, waist circumference, blood pressure, skeletal muscle mass, and omega index
* Psychiatric symptom measures include: mood, psychosis, cognition, and quality of life
* Deep omic profiling including metabolic and proteomic data. Through identifying patterns, changes, and pathways of molecular, psychiatric, physiologic, and metabolic markers, the investigators aim to assess how this intervention may impact individuals with serious mental illnesses and symptoms/conditions related to serious mental illnesses.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with bipolar disorder (BD), major depressive disorder (MDD), and or schizophrenia

   1. For individuals diagnosed with bipolar disorder (BD):

      * Meet DSM V criteria for BD (any subtype)
      * Not mild
      * >40 on BPRS
      * clinically stable (with no hospitalization for past 3 months)
   2. For individuals diagnosed with major depressive disorder (MDD):

      * Not mild
      * PHQ-9 > 10
      * clinically stable (with no hospitalization for past 3 months)
   3. For individuals diagnosed with schizophrenia:

      * Meet DSM V criteria for schizophrenia (any subtype)
      * Not mild
      * >40 on BPRS
      * clinically stable (with no hospitalization for past 3 months)
2. Participants may currently be on a stable and adequate dose of SSRI antidepressant therapy or other psychiatric medication. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, or trazodone) will be allowed if the therapy has been stable for at least four weeks prior to screening and if it is expected to remain stable. Participants may be switched from other classes of medication to another medication class by their psychiatrist or primary care doctor, but need to be stable enough to enroll and adhere to study procedures.
3. willing and able to give informed consent for participation in English.
4. live within the United States.

   --------------------------------------------------------------------------------

Exclusion Criteria:

1. has started the ketogenic diet or was in ketosis within 3 months of wanting to enroll
2. pregnant or nursing
3. insulin dependent
4. comorbidity of developmental delay
5. in a current severe mood or psychotic state when entering the study that would prohibit compliance with study visits or dietary programs.
6. any one who has been hospitalized or taken clozapine at doses above 550mg over the past 3 months
7. inability to complete baseline measurements
8. severe renal or hepatic insufficiency
9. cardiovascular dysfunction, including diagnosis of:

   * Congestive heart failure
   * Angina
   * Arrhythmias
   * Cardiomyopathy
   * Valvular heart disease
10. active substance abuse with illicit drugs or alcohol and/or current diagnosis of a Substance Use Disorder (Abuse or Dependence, as defined by DSM-IV-TR), with the exception of nicotine or cannabis dependence
11. active suicidal and considered at significant risk for suicide during course of study
12. participation in any clinical trial- within the past month or concurrent to study participation- with an investigational drug/device and/or intervention that may interfere with study participation/evaluation of results
13. mild BPRS at screening or baseline visits
14. history of TBI
15. any other medical condition that may make diet intervention dangerous as determined by the study medical team (e.g. anorexia nervosa) or assessed by study team to have insufficient control over their food intake to adhere to study diets.
16. any medical condition that physicians or the PI believe would interfere with study participation or evaluation of results
17. history of familial hypercholesterolemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
WHO-5 Well-being Index | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in general well-being from baseline. Self reported to measure quality of life. Assessed on 5-items, scored from 0-5 on each item, with higher scores indicating better quality of life.
Functioning Assessment Short Test (FAST) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in quality of life from baseline. Self reported and assessed on 24-items regarding difficulties in the experiences described. Scored from 0-3 on each item, with lower composite scores indicating better quality of life.
Quality of Life Scale (QIDS) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in severity of depression from baseline. Self reported on 16 items with a composite score range of 0-27 (0= no depression, 27 = very severe depression).

SECONDARY OUTCOMES:
Cambridge Cognition (CANTAB Assessment) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in cognition and brain health assessment from baseline. Scored by assessment's algorithm that compares scores within the established benchmark by age group and test. (≥ 1.5 SD below normative means = insufficient performance, ≥1 SD below normative means = subtle impaired performance in task)
Quality of Life in Neurological Disorders (Neuro-QOL, Cognitive Function) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in quality of life related to cognitive function from baseline. T-score 17.3- 38.9 (high scores indicate better/desirable self-reported health).
Brief Psychiatric Assessment Scale (BPRS) | Screening; Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  change in severity of psychopathy; 18 conditions scored by clinician. Each of the 18 conditions/outcomes rated from 0-7 (0= not assessed, 7 = extremely severe).
Patient Health Questionnaire (PHQ-9) | Screening; Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in Depression; 9-10 items scored on composite score range 0-27 (0= no depression, 27= severe depression).
Clinical Global Impressions Scale (CGI)/ Clinical Mood Monitoring | Screening; Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in Clinical Global Impression (CGI) Psychiatric Index; 1-7 scale. (1= not at all ill, 7= among the most extremely ill patients).
Perceived Stress Scale 4 (PSS-4) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in perceived stress from baseline measured by PSS-4 biweekly, a 4-item scale providing a 0-16 point composite score, with higher scores indicating greater perceived stress.
Generalized Anxiety Disorder Scale (GAD-7) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in General Anxiety Disorder (GAD-7) scale from Baseline. 0-15+ scale. (0= no anxiety, 15+= severe anxiety).
Pittsburgh Sleep Quality Index (PSQI) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in sleep quality from baseline; 0-21 scale (<5=good sleeper; 5+= meaningfully disturbed sleep or poor sleeper).
Epigenome | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Profiling of epigenome measured in biospecimen collected.
Mitochondrial Function | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in mitochondrial function from baseline measured in biospecimen.
Metabolome | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in metabolites from baseline measured in biospecimen.
Proteome | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in proteins from baseline measured in biospecimen.
Microbiome | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in microbes/microorganisms from baseline measured in biospecimen.
Transcriptome | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in mRNA-based expression from baseline measured in biospecimen.
Lipidome | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in lipids from baseline measured in biospecimen.
Blood pressure | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in blood pressure measured continuously by wearable devices and recorded weekly/biweekly during study visits.
Heart Rate Variability | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in heart rate variability measured continuously by wearable devices and recorded weekly/biweekly during study visits.
Heart Rate | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in heart rate measured continuously by wearable devices and recorded. weekly/biweekly during study visits.
Weight | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in Weight from Baseline, recorded weekly/biweekly during study visits.
Waist Circumference | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Change in waist circumference from Baseline, recorded weekly/biweekly during study visits.
Total Cholesterol | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Blood measurement of change in Lipid Profile (total cholesterol) from baseline.
Low Density Lipoprotein Cholesterol (LDL-C) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Blood measurement of change in Lipid Profile (LDL-C) from baseline.
High Density Lipoprotein Cholesterol (HDL-C) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Blood measurement of change in Lipid Profile (HDL-C) from baseline.
Triglycerides (TG) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Blood measurement of change in Lipid Profile (TG) from baseline.
Inflammatory Marker (hs-CRP) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Blood measurement of change in Inflammatory Marker (hs-CRP) from baseline.
Insulin Resistance Measure (HOMA-IR) | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Blood measurement of change in insulin resistance from baseline.
Glucose | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Blood measurement of change in Metabolic Marker (Glucose) from baseline.
Hemoglobin A1c | Baseline through study completion, an average of 12 weeks (Arm 1: Ketogenic Diet Only) or 24 weeks (Arm 2: DAU-Ketogenic Diet Crossover).
  Blood measurement of change in Metabolic Marker (hemoglobin A1c) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Shebani Sethi, MD, ABOM, Principal Investigator — Stanford University; Michael Snyder, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

REFERENCES:
- [Background] Leucht S, Kane JM, Kissling W, Hamann J, Etschel E, Engel R. Clinical implications of Brief Psychiatric Rating Scale scores. Br J Psychiatry. 2005 Oct;187:366-71. doi: 10.1192/bjp.187.4.366. PMID 16199797